CLINICAL TRIAL: NCT04041843
Title: A Pilot Study of an Oral Anticoagulant "Apixaban" for theTreatment of Venous Thromboembolism in Children and Adolescents
Brief Title: Oral Anticoagulant Apixaban for Treatment of Venous Thromboembolism
Acronym: VTE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYMC 191
Record Dates: First submitted 2019-07-31; First posted 2019-08-01 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Abixaban (Experimental): Apixaban 10 mg twice daily p.o. for seven days followed by 5 mg twice daily p.o. for children and adolescents weighting ≥40 kg who have been diagnosed with a thrombosis.
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban — Apixaban 10 mg twice daily p.o. for seven days followed by 5 mg twice daily p.o. for children and adolescents weighting ≥40 kg
  Other Names: Eliquis

SUMMARY:
Patients who have developed a venous thrombosis will receive apixaban to treat and prevent a secondary thromboembolism.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents with a newly diagnosed primary VTE.
* Treatment with apixaban has to begin within 72 hours of the diagnosis of VTE.
* Patients who have received heparin at the beginning of their diagnosis and are willing to switch to apixaban, are allowed to do so within 72 hours of their treatment. Patients who are switched to apixaban are not allowed to receive any other systemic anticoagulant therapy.
* VTE confirmed by diagnostic imaging.
* Children with body weight of ≥ 40 kg and are able to tolerate medication by mouth or administered via an NG or GT tube.
* Adequate liver function: AST and/or ALT <5 times ULN, and/or Direct bilirubin <2 times ULN
* Platelet count of at least ≥ 30,000/ul.
* Adequate renal function: >30% of GFR for age
* Female subjects of childbearing potential must not be nursing or pregnant with negative urine pregnancy test within 72 hours prior to dosing with study medication.
* Signed written informed consent

Exclusion Criteria:

* Current or recent (within 3 months) apixaban administration.
* Patient is unable to tolerate medications by oral route or by n/g administration, peptic ulcer disease, intestinal obstruction, toxic megacolon, typhlitis, or short gut syndrome.
* History of primary bleeding disorder and first degree family history of bleeding disorder.
* Active bleeding or high risk of bleeding at the time of study entry.
* History of significant head injury and/or any history of intracranial hemorrhage.
* Conditions predispose to intracranial bleed; e.g. brain tumor, brain metastasis.
* Uncontrolled Grade 3 or 4 severe hypertension.
* History of allergy to apixaban or factor Xa inhibitors.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
venous thromboembolism (VTE) formation | 7-90 days
  No new VTE

SECONDARY OUTCOMES:
Doppler ultrasound vein imaging | day 8-15
  Change in VTE on Doppler ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Oya Tugal, MD, Principal Investigator — New York Medical College
Locations (1):
- New York Medical College, Valhalla, New York, United States